CLINICAL TRIAL: NCT00663728
Title: A Randomized, Double-blind, Crossover Study to Evaluate the Duration of Erection Following Vardenafil (10mg) Administration for Four Weeks in a Fixed Dose Regimen Compared to Placebo in Males With ED
Brief Title: Assessment of Duration of Erection With Vardenafil 10 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11575
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10mg Vardenafil taken orally 1 hour prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
This study assessed the effect of 10mg vardenafil, taken on demand in an 'at home' setting, as compared to placebo (dummy medication with no pharmacological activity), on the duration of erection from the moment when the patient perceived his erection to be hard enough for penetration until withdrawal from the partner's vagina leading to successful completion which may or may not have included ejaculation. The patient used the stopwatch for the above assessments. The efficacy of oral ED treatments is measured by questionnaires and patient diaries.

ELIGIBILITY:
Inclusion Criteria:- Males with erectile dysfunction- Stable heterosexual relationship Exclusion Criteria:- Primary hypoactive sexual desire- History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months nitrate use

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2004-09; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Effect of vardenafil on the duration of erection | 4 weeks

SECONDARY OUTCOMES:
Perception of erection to be hard enough for penetration | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer